CLINICAL TRIAL: NCT00005323
Title: Epidemiology of Persistent Pulmonary Hypertension of the Newborn - SCOR in Lung Biology and Diseases in Infants and Children
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4104; P50HL046491 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2001-10

CONDITIONS: Lung Diseases; Cardiovascular Diseases; Defect, Congenital Heart; Heart Diseases; Persistent Fetal Circulation Syndrome
MeSH Terms: conditions — Lung Diseases; Cardiovascular Diseases; Heart Defects, Congenital; Heart Diseases; Persistent Fetal Circulation Syndrome

SUMMARY:
To conduct an epidemiologic study of persistent pulmonary hypertension of the newborn ( PPHN) infant.

DETAILED DESCRIPTION:
BACKGROUND:

The study on the epidemiology of persistent pulmonary hypertension of the newborn (PPHN) was a subproject within a Specialized Center of Research (SCOR) in Lung Biology and Diseases in Infants and Children. The SCOR and its subproject were awarded in December, 1991. Dollars were estimated at 20 percent of total center dollars.

DESIGN NARRATIVE:

Data from a previous study of PPHN were analyzed. The objectives were to: identify the effects of a variety of potentially adverse prenatal exposures from interview data; formulate multi-variate models of risk of PPHN to determine if smoking or use of prostaglandin inhibitors increased the risk of PPHN; explore associations of PPHN with history of illicit drug use and maternal hypoxia; examine the relationships of postnatal care and perinatal risk factors on the incidence and outcome of PPHN; test the relationships of PPHN to the biochemical presence of nicotine and drugs in neonatal urine.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-12; Study Completion 1996-11 (Actual)

REFERENCES:
- [Background] Derkach IuS, Osherovich AM, Miasnenko AM. [Organization of the equipment and public health measures in virological laboratories of epidemiological health stations]. Lab Delo. 1984;(6):374-7. No abstract available. Russian. PMID 6206298
- [Background] Christou H, Adatia I, Van Marter LJ, Kane JW, Thompson JE, Stark AR, Wessel DL, Kourembanas S. Effect of inhaled nitric oxide on endothelin-1 and cyclic guanosine 5'-monophosphate plasma concentrations in newborn infants with persistent pulmonary hypertension. J Pediatr. 1997 Apr;130(4):603-11. doi: 10.1016/s0022-3476(97)70245-2. PMID 9108859